CLINICAL TRIAL: NCT05420727
Title: Theranostics in Soft Tissue Sarcoma Using a Vascular Disruption Approach
Acronym: ThernSarc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John O. Prior (Other)
Responsible Party: Sponsor-Investigator, John O. Prior, Head of Nuclear Medicine Department, PhD MD, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Theranostics STS
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Ga-68-PSMA-11 PET/CT patients treated by Lu-177-ITG-PSMA-1 (Experimental): Positive Ga-68-PSMA-11 PET/CT prior to two cycles of Lu-177-ITG-PSMA-1 i scheduled six weeks apart.
  Interventions: Drug: Ga-68-PSMA-11 PET/CT; Drug: Lu-177-ITG-PSMA-1

INTERVENTIONS:
Drug: Ga-68-PSMA-11 PET/CT — Ga-68-PSMA-11 PET/CT imaging
Drug: Lu-177-ITG-PSMA-1 — Lu-177-ITG-PSMA-1 treatment

SUMMARY:
To test the feasibility of theranostic targeting the PSMA receptor in STS patients by Ga-68-PSMA-11 PET/CT and Lu-177-ITG-PSMA-1 treat-ment with special emphasis on vascular disruption using a translational approach.

ELIGIBILITY:
Inclusion Criteria:

* Female or male ≥ 18 years old at the time of informed consent
* Patients with proven Soft Tissue Sarcoma
* Patients need to pass the sarcoma tumor board and the molecular tumor board at CHUV and no approved therapeutic alternative is available
* Progression of the disease by RECIST v1.1 after standard therapies according to the treat-ing oncologists
* Informed Consent as documented by signed informed consent form

Exclusion Criteria:

* Patients under active anti-sarcoma treatment other than the study product (Lu-177-ITG-PSMA-1)
* Female participants who are pregnant or breast feeding
* Female participants with intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not us-ing and not willing to continue using a medically reliable method of contraception for the en-tire study duration until 6 months after last Lu-177-ITG-PSMA-1 treatment, such as oral, in-jectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Male patients of reproductive potential, not using and not willing to use a medically reliable method of contraception for the entire study duration until 6 months after last Lu-177-ITG-PSMA-1 treatment, such as barrier method or sexual abstinence or who are not using any other method considered sufficiently reliable by the investigator in individual cases. The par-ticipant must inform their female partners about the participation in this trial and they must use additional effective contraception (e.g., hormonal) during the trial until 6 months after the last Lu-177-ITG-PSMA-1 treatment.
* Previous enrolment into the current study
* History of any disease or relevant physical condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment
* Insufficient knowledge of project language, inability to give consent or to follow procedures, incapacity to follow radiation safety procedures, required by the study
* Enrolment of the investigator, his/her family members, employees and other dependent per-sons
* The patient makes use of his/her "right not to know" and refuses to be informed about inci-dental findings
* Absence of PSMA accumulation in at least 50% of tumours on Ga-68-PSMA-11 PET/CT
* Grade IV renal impairment and above (calculated GFR < 30 mL/min/1.73 m2)
* Blood count disturbance:

Platelets < 75,000/µL. Leukocytes < 2,500/µL Haemoglobin < 80 g/L. • Disturbance of liver function with: Total bilirubin > 2 times the upper limit of the norm ASAT/ALAT > 3 times the upper limit without the presence of liver metastases ASAT/ALAT > 5 times the upper limit in the presence of liver metastases

• Hypersensitivity to any of the ingredients of the injectable product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
imaging result obtained by Ga-68-PSMA-11 PET/CT | four weeks after the second cycle of Lu-177-ITG-PSMA-1 treatment, compared to base-line

SECONDARY OUTCOMES:
SUVmax and radiological changes using PSMA - PET/CT | four weeks after the second cycle of Lu-177-ITG-PSMA-1 treatment, compared to base-line.
  SUVmax and radiological changes using PSMA - PET/CT using advanced radiological assessment including CHOI criteria to as-sess the necrosis one month after end of second cycle
Tumor evaluation using contrast enhanced computed tomography (ceCT) | four weeks after the second cycle of Lu-177-ITG-PSMA-1 treatment, compared to base-line.
  Tumor evaluation using contrast enhanced computed tomography (ceCT) using RECIST v1.1 (change in tumor size in mm)

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois - Lausanne University Hospital
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No